CLINICAL TRIAL: NCT04813757
Title: Scapular Upward Rotation Focused Treatment for Patients With Shoulder Impingement Syndrome and a Positive Scapular Assistance Test
Brief Title: Scapular Upward Rotation Focused Treatment for Patient With Shoulder Impingement Syndrome and a Positive Scapular Assistance Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meuhedet. Healthcare Organization (Other)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-06-11-19
Record Dates: First submitted 2020-12-20; First posted 2021-03-24 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Subacromial Pain Syndrome; Impingement Syndrome; Scapular Dyskinesis
MeSH Terms: interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: We assume participants will not be able to differentiate between the upward rotation focused intervention and the control intervention. Furthermore, the examiner performing baseline and outcome assessment will be unaware of the group allocation while performing these assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group will receive 12 treatment sessions over a 6-week period. Three sessions during the first 2 weeks, 2 sessions per week during weeks 3 and 4 , and one session during weeks 5 and 6. Each session will be 30 minutes including 10 minutes of manual therapy and 20 minutes for review and/or modification of the exercise program. The manual therapy will include trigger point manual therapy. The exercise program will include 2 scapular and rotator cuff strengthening exercises emphasizing scapular upward rotation and posterior tilt and one additional flexibility exercise. These exercise will be repeated at home on the days in between the therapy sessions.
  Interventions: Other: exercise; Other: manual therapy
- control group (Active Comparator): Participants in the control group will receive 12 treatment sessions over a 6-week period. Three sessions during the first 2 weeks, 2 sessions per week during weeks 3 and 4 , and one session during weeks 5 and 6. Each session will be 30 minutes including 10 minutes of manual therapy and 20 minutes for review and/or modification of the exercise program. The manual therapy will include trigger point manual therapy, posterior shoulder stretching, and mobilization-with-movement into shoulder elevation. The exercise program will include 2 exercises focusing on scapular and rotator cuff strengthening without a special emphasis on scapular upward rotation as well as one additional flexibility exercise. These exercises will be performed at home on the days on between the therapy sessions.
  Interventions: Other: exercise; Other: manual therapy

INTERVENTIONS:
Other: exercise — each group will perform 2 shoulder strength exercise at the therapy session and 3 exercise at home session-2 strength exercise and one stretching exercise. they will perform the exercises 5 times per week
Other: manual therapy — on each treatment session both group will receive 15 minutes of manual therapy which will include: massage,3-4 trigger point treatment posterior capsule stretch and mobilization with movement

SUMMARY:
Altered scapular movement is a common impairment among patients with subacromial impingement syndrome (SAIS). Nevertheless scapular focused interventions have resulted in conflicting findings among this population. One possible reason for this is the inability to identify patients with SAIS who will respond favorably to a scapular focused intervention.

The scapular assistance test (SAT) may be one possible indicator of patients most likely to benefit from a scapular focused intervention, particularly one that emphasizes scapular upward rotation. The purpose of this study is to examine targeted upward rotation intervention in patients demonstrating a positive Scapular Assistance test.

DETAILED DESCRIPTION:
Background: Patients with SAIS are commonly referred to physical therapy. A common impairment among patients with SAIS is altered scapular movement, characterized by insufficient upward rotation and posterior tilt. These deficits are believed to decrease the subacromial space and diminish length -tension relationship among the deltoid and rotator cuff musculature. The scapular assistance test (SAT) is a physical examination manoeuvre aimed to detect patients in whom insufficient scapular upward rotation and posterior tilt contribute to the generation of shoulder symptoms. The SAT may, therefore, serve as an indication for the need of scapular focused intervention. Given the inconsistent results of scapular focused interventions among patients with SAIS, the purpose of this study is to assess the outcome of a scapular-focused intervention, particularly geared toward increasing scapular upward rotation, among patients with SAIS that exhibit a positive SAT as well.

Methods: Fifty patients with SAIS and a positive SAT referred to the "Meuhedet" outpatient physical therapy clinic in Ashdod will be recruited for this study. Following baseline assessment, patients will be randomized into 12 sessions over a 6-week period. The intervention group will receive manual therapy and an exercise program focused on increasing scapular upward rotation while the control group will receive manual therapy and an exercise program focused on scapular muscle an rotator cuff strengthening with no special emphasis on scapular upward rotation. Repeated measures analysis of covariance will be conducted to detect differences in pain intensity, shoulder -related disability and scapular upward rotation following the intervention

ELIGIBILITY:
Inclusion Criteria:

* Unilateral shoulder pain for ≥1 month
* A diagnosis of SAIS as determined by having 3 or ore positive tests out of: Neer test, Hawkins test, Painful arc, Jobe test, external rotation resistance test.
* A positive SAT

Exclusion criteria:

* Cervical spine involvement as evidenced by reproduction of symptoms with neck movement
* Massive rotator cuff tear as evidenced by pseudoparalysis
* Previous history of a fracture or surgery within the involved shoulder.
* Limited passive range of motion by ≥50% or more compared with uninvolved side in

  * 2 planes of motion (i.e. flexion, external rotation)
* A history of shoulder dislocation or subluxation
* A history of Rheumatoid arthritis, CVA, fibromyalgia
* Current pregnancy
* Population with special needs
* Pending disability claim / litigation procedure associated with shoulder complaint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disability of the Arm, Shoulder and Hand (DASH) questionnaire | pre intervention
  each participant will receive the Disability of the Arm shoulder and hand questioner. score is from 0 -100 a higher score is greater disability
Numeric pain Rating Scale (NPRS), 0 - 10 | pre intervention
  each participant will receive the NPRS questioner higher score means greater pain

SECONDARY OUTCOMES:
Active shoulder flexion | pre intervention
  in standing position the patient will elevate the arm in the sagittal plane, the range of motion will be measured by goniometer
active shoulder abduction | pre intervention
  in standing position the patient will elevate the arm in the frontal plane, the range of motion will be measured by goniometer
scapular posterior tilt | pre intervention
  in standing position the scapular posterior tilt willl be measured by digital inclinometer which will be placed on the medial border of the scapula. the posterior tilt will be measured in 90 and 120 degree of forward flexion

CONTACTS AND LOCATIONS:
Locations (1):
- Meuhedet, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No